CLINICAL TRIAL: NCT02262806
Title: Compassionate Use of Metreleptin in Previously-Treated Patients With Partial Lipodystrophy
Brief Title: Compassionate Use of Metreleptin in Previously Treated People With Partial Lipodystrophy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150002; 15-DK-0002
Record Dates: First submitted 2014-10-09; First posted 2014-10-13 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-11-20

CONDITIONS: Diabetes; Lipodystrophy; Hyperlipidemia
Keywords: Lipodystrophy; Leptin; Hypertriglyceridemia; Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Lipodystrophy; Hyperlipidemias; Hypertriglyceridemia | interventions — metreleptin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Leptin therapy (Other): leptin administered via SC injections BID
  Interventions: Drug: Metreleptin

INTERVENTIONS:
Drug: Metreleptin — A leptin analog indicated as an adjunct to diet as replacement therapy to treat the complications of leptin deficiency in patients with partial lipodystrophy.

SUMMARY:
Background:

- Partial lipodystrophy can cause high blood fat levels and resistance to insulin. This can lead to health problems including diabetes. Researchers have found that the drug metreleptin improves health in people with this disease.

Objective:

- To test the safety and effectiveness of metreleptin.

Eligibility:

* People age 6 months and older with partial lipodystrophy who
* have received metreleptin through NIH studies and shown improvement AND
* cannot get metreleptin other ways.

Design:

* Participants will come to NIH approximately every 6 months during year one, then every 1 2 years. Financial assistance may be available for travel within the U.S.
* At visits, participants will get a supply of metreleptin to take home for daily injections, or it can be shipped to them inside the U.S. They will have:
* plastic catheter placed in an arm vein.
* blood tests, urine collection, and physical exam.
* oral glucose tolerance test, drinking a sweet liquid.
* ultrasound of the heart, liver, uterus, and ovaries. A gel and a probe are placed on the skin and pictures are taken of the organs.
* echocardiogram, which takes pictures of the heart with sound waves.
* Resting Metabolic Rate taken. A plastic hood is worn over the head while the oxygen they breathe is measured.
* Participants will have up to 3 DEXA scan x-rays per year.
* Participants may have:
* annual bone x-rays.
* liver biopsies every few years. A needle will be inserted into the liver to obtain a small piece. Participants will sign a separate consent for this.
* Participants must be seen regularly by their local doctors and have blood tests at least every 3-6 months at home.

DETAILED DESCRIPTION:
Leptin is an adipocyte-derived hormone that can be thought of as a signal from adipose tissue to the rest of the body conveying information about long-term nutritional status. Patients with lipodystrophy have leptin deficiency secondary to lack of adipose tissue. The combination of leptin deficiency and ectopic lipid deposition in patients with lipodystrophy leads to metabolic complications including severe insulin resistance and diabetes, hypertriglyceridemia, non-alcoholic steatohepatitis, and polycystic ovarian syndrome. Between 2000 and 2014, the NIDDK IRP conducted an open-label clinical trial of the recombinant human leptin analog, metreleptin, in patients with generalized and partial forms of lipodystrophy. This study showed that metreleptin ameliorates metabolic and endocrine abnormalities in lipodystrophy, including reducing food intake, improving insulin resistance and diabetes, reducing ectopic lipid, and normalizing reproduction. Based on these data, metreleptin was approved by the FDA in February, 2014, for patients with generalized, but not partial, lipodystrophy. Our data have shown, however, that a subgroup of patients with partial lipodystrophy do gain medical benefit from metreleptin.

The purpose of this study is twofold:

* To provide access to metreleptin to patients with partial lipodystrophy who have previously received and derived benefit from metreleptin through NIH studies (protocols 02-DK-0022 and 13-DK-0057).
* To continue to collect data on the long-term efficacy of metreleptin in ameliorating the metabolic complications of partial lipodystrophy.

Metreleptin will be given at doses of less than or equal to 0.24 mg/kg/day, adjusted based on body weight and metabolic control. Patients will be seen approximately once per year at NIH for evaluation, and potentially less frequently for those who are medically stable and have difficulty traveling to NIH. Laboratory evaluation will be obtained more frequently by the patient s home providers as clinically indicated. The primary outcomes of the study are improvements in serum triglycerides and hemoglobin A1c levels. Secondary outcomes include measures of steatohepatitis and ectopic lipid, body composition, bone mineral density and bone mineral metabolism, and pituitary and reproductive function.

Metreleptin is supplied by Chiesi USA, Inc. Neither the NIH nor Chiesi USA, Inc. can guarantee that leptin will be available indefinitely and/or after the study ends.

ELIGIBILITY:
* INCLUSION CRITERIA
* Age greater than or equal to 6 months
* Partial lipodystrophy (either genetic or acquired)
* Previously or currently treated with metreleptin under NIH study 02-DK-0022 and/or NIH study 13-DK-0057.
* Documented metabolic benefit from prior or current metreleptin treatment, defined as one or more of the following:

  * TG reduction greater than or equal to 30% OR
  * HbA1c reduction greater than or equal to 1% OR
  * Decrease in insulin requirements greater than or equal to 40% OR
  * Decrease in episodes of pancreatitis OR
  * Improvement in steatohepatitis OR
  * Withdrawal of metreleptin led to marked worsening of metabolic parameters

EXCLUSION CRITERIA

* Availability of metreleptin to the patient either as an approved drug, or through local compassionate use or expanded access programs.
* Known HIV infection or HIV-associated lipodystrophy.
* Psychiatric disorder impeding competence or compliance.
* Any medical condition or medication that will increase risk to the subject.
* Current alcohol or substance abuse.
* Subjects who have a known hypersensitivity to E. coli derived proteins.

Ages: 6 Months to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-10-14 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Serum hemoglobin A1C | every 6-12 months
  improvement in lab value
Serum triglycerides | every 6-12 months
  improvement in lab value

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca J Brown, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Subject level data will be shared upon request after appropriate collaboration agreements are in place.

REFERENCES:
- [Background] Akinci B, Oral EA, Neidert A, Rus D, Cheng WY, Thompson-Leduc P, Cheung HC, Bradt P, Foss de Freitas MC, Montenegro RM, Fernandes VO, Cochran E, Brown RJ. Comorbidities and Survival in Patients With Lipodystrophy: An International Chart Review Study. J Clin Endocrinol Metab. 2019 Nov 1;104(11):5120-5135. doi: 10.1210/jc.2018-02730. PMID 31314093
- [Derived] Sekizkardes H, Cochran E, Malandrino N, Garg A, Brown RJ. Efficacy of Metreleptin Treatment in Familial Partial Lipodystrophy Due to PPARG vs LMNA Pathogenic Variants. J Clin Endocrinol Metab. 2019 Aug 1;104(8):3068-3076. doi: 10.1210/jc.2018-02787. PMID 31194872
- [Derived] Brown RJ, Meehan CA, Cochran E, Rother KI, Kleiner DE, Walter M, Gorden P. Effects of Metreleptin in Pediatric Patients With Lipodystrophy. J Clin Endocrinol Metab. 2017 May 1;102(5):1511-1519. doi: 10.1210/jc.2016-3628. PMID 28324110
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-DK-0002.html